# REPUBLIC OF TURKIYE ANKARA YILDIRIM BEYAZIT UNIVERSITY INSTITUTE OF HEALTH SCIENCES

## "EVALUATION OF THE EFFECT OF PENDER'S HEALTH PROMOTION THEORY BASED DIABETES SELF-MANAGEMENT PROGRAM ON HEALTHY LIVING BEHAVIORS IN PREGNANT WOMEN DIAGNOSED WITH GESTATIONAL DIABETES MELLITUS"

INFORMED CONSENT FORM FOR PREGNANT WOMEN IN THE INTERVENTION GROUP

#### **INFORMED CONSENT FORM**

#### PLEASE TAKE TIME TO READ THIS DOCUMENT CAREFULLY

We invite you to the study titled "Evaluation of the Effect of Pender's Health Promotion Theory Based Diabetes Self-Management Program on Healthy Living Behaviors in Pregnant Women Diagnosed with Gestational Diabetes Mellitus" conducted by Specialist Nurse Esra ALTUN under the supervision of Prof. Dr. Sena KAPLAN. Before deciding whether to participate in this study, you need to know why and how the study will be conducted. Therefore, it is very important to read and understand this form. If there is anything you do not understand or that is not clear to you, or if you want more information, please ask us.

Participation in this study is completely voluntary. You have the right not to participate in the study or to withdraw from the study at any time after participating. Your response to the study will be interpreted as your consent to participate in the study. Do not be under pressure or suggestion from anyone while answering the questions on the forms given to you. The information obtained from these forms will be used solely for research purposes.

- 1. Information Related to the Research:
- a. Purpose of the Research: It is aimed to evaluate the effect of the nursing education intervention prepared based on the health promotion model for pregnant women diagnosed with gestational diabetes on gestational diabetes management and healthy lifestyle behaviors.
- b. Content of the Research: Data will be collected from the participants with the Personal Information Form, Healthy Lifestyle Behaviors (HLB) Scale II, Self-Efficacy Scale in Gestational Diabetes, Health Belief Model Scale in Diabetic Patients, Multidimensional Perceived Social Support Scale.
- c. Reason for the Research: Thesis study
- d. Estimated Duration of the Research: The survey application time is planned as 20 minutes on average.
- e. Number of Participants/Volunteers Expected to Participate in the Research: 68

| f. | Place | of | Study: | Ankara | University | Health | Practice | and | Research | Hospitals, | Department | of |
|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Obstetrics and Gynecology | | | | | | | | | | | | |

### 2. Consent to Participate in the Study:

Signature:

I have read the information provided above that should be given to the participant/volunteer before the study and I fully understand the scope and purpose of the study in which I am asked to participate and the responsibilities that fall upon me as a volunteer. Written and verbal explanations about the study were made by the researcher named below, I had the opportunity to ask questions and discuss and received satisfactory answers. The possible risks and benefits of the study were also explained to me verbally. I understand that I can leave this study at any time and without having to state any reason and that I will not encounter any negative consequences if I do so.

| Under these conditions, I agree to participate in the study of my own free will, without any pressure or |
|---|
| coercion. |
| Name-Surname: |